CLINICAL TRIAL: NCT06651814
Title: Treatment Outcome of Supervised Exercise and Home Exercise in Patients with Symptomatic Disc Displacement with Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Armed Forces Institute of Dentistry, Pakistan (Other)
Responsible Party: Principal Investigator, Dr. Ayesha Younas, Principal Investigator, Armed Forces Institute of Dentistry, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AYounas
Record Dates: First submitted 2024-10-17; First posted 2024-10-22 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Anterior Disc Displacement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Supervised Exercise Group (Experimental): Patients receive supervised exercise therapy from a qualified physical therapist or healthcare professional, with a set frequency and duration
  Interventions: Behavioral: Supervised Exercise Group
- Home Exercise Group (Active Comparator): Patients receive written instructions and demonstrations for performing exercises at home, with recommended frequency and duration
  Interventions: Behavioral: Home Exercise Group

INTERVENTIONS:
Behavioral: Supervised Exercise Group — A supervised exercise program will consists of 10 sessions. The 1st exercise station will be a 5-minute warming up of the jaw with a heat lamp. The 2nd station will involve jaw opening-closing movements (TMJ rotation) with the mandible in a slightly protruded position for 6 minutes. The 3rd and 4th exercise stations will comprised of jaw opening and jaw protrusion, respectively, against resistance for 4 minutes each. Measurements will be done before the trial started and after 3 months.
  Arms: Supervised Exercise Group
Behavioral: Home Exercise Group — Patients will received a home regime of jaw exercises. They will be instructed to do two different trainings. The 1st type of exercise will be jaw opening and closing movements daily for 5 minutes after each meal with the mandible and the head of the TMJ in a slightly protruded position. This exercise should not produce any clicking sounds. The 2nd type of exercise will be isometric exercises; this entailed jaw opening and jaw protrusion against resistance with their hand for 10 seconds with 10 repetitions each daily. All the patients will receive a training brochure with photos of the exercises and detailed information on frequency and exercise time. The brochure will include a diary. After 6 weeks, the subject and the assistant will check the performance of the exercise and the diary
  Arms: Home Exercise Group

SUMMARY:
The aim of the study is to evaluate the treatment outcome of supervised exercise and home exercise in patients with symptomatic disc displacement with reduction.

DETAILED DESCRIPTION:
This study will help the clinical practitioner to choose better exercise option in patients with symptomatic disc displacement with reduction in order to avoid clicking sound.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70 years
2. Both genders
3. TMJ clicking sounds fulfilling RDC/TMD for symptomatic disc displacement

   1. Clicking sounds during jaw opening and closing
   2. Interincisor distance ≥ 5mm wider during mouth opening
   3. Clicking suppression with protruded mandible
   4. Clicking presence in at least two of three repetitions
4. NRS score ≥ 4 for TMJ clicking sound severity
5. TMJ clicking sound frequency: once a week or more

Exclusion Criteria:

1. Major psychiatric disorders
2. Ongoing treatments related to symptoms
3. Active rheumatologic disease
4. Malignant disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
clicking sounds frequency | 3 months
  Assessment of clicking sounds frequency before and after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Younas, BDS, Principal Investigator — Armed Forces Institute of Dentistry, Pakistan
Locations (1):
- Armed Forces Institute of Dentistry, Rawalpindi, Punjab Province, Pakistan